CLINICAL TRIAL: NCT01052454
Title: Pilot Study to Assess the Feasibility of MBSR for Hot Flashes
Brief Title: Mindfulness-Based Stress Reduction for Hot Flashes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: James Carmody, University of Massachusetts Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT002910
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Vasomotor Symptoms
Keywords: hot flashes; mindfulness; stress
MeSH Terms: conditions — Hot Flashes | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait list (No Intervention): Women assigned to the waitlist have the opportunity of taking the MBSR program at no cost following final study assessment
- Mindfulness-based stress reduction (Experimental): Women in the MBSR arm attend eight weekly MBSR classes
  Interventions: Behavioral: Mindfulness-based stress reduction

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction — Participants in the MBSR arm attend eight weekly classes.
  Other Names: MBSR
  Arms: Mindfulness-based stress reduction

SUMMARY:
This is a study to determine if participation in a mindfulness-based stress reduction program is feasible for women experiencing five or more hot flashes/day, and whether it affects either the frequency and/or intensity of their hot flashes, or the degree of bother they experience from them

ELIGIBILITY:
Inclusion Criteria:

* Women experiencing 5 or more hot flashes/day

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-09; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Hot Flash intensity/bother

CONTACTS AND LOCATIONS:
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States